CLINICAL TRIAL: NCT06751563
Title: A Randomized Pilot Study of Produce Prescription Programs in Adults With Overweight or Obesity Experiencing Nutrition Insecurity
Brief Title: Study of Produce Prescription Programs in Adults With Overweight or Obesity Experiencing Nutrition Insecurity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Maryland Department of Health and Mental Hygiene (Other Government); Maryland Cigarette Restitution Fund (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00463007
Record Dates: First submitted 2024-12-20; First posted 2024-12-30 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Overweight and Obesity
Keywords: obesity; overweight; produce prescription; produce voucher; nutrition; nutrition security
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Produce Voucher (Experimental): Behavioral Text Message Program + Produce Voucher
  Interventions: Behavioral: Behavioral Text Message Program and Produce Voucher
- Produce Boxes (Experimental): Behavioral Text Message Program + Produce Box Delivery
  Interventions: Behavioral: Behavioral Text Messages and Produce Box Delivery

INTERVENTIONS:
Behavioral: Behavioral Text Messages and Produce Box Delivery — Participants will receive a produce box delivered weekly to the participants home customized based on the participants cooking preferences and household size. Participants will also receive a daily text message aimed to support a healthy diet and lifestyle. These texts will include information to build participants' knowledge and skills for healthy eating. The participants will also include weekly goals that focus on eating a healthy diet. Participants will receive automated, personalized feedback via text messages based on participant goal attainment and daily responses.
  Arms: Produce Boxes
Behavioral: Behavioral Text Message Program and Produce Voucher — Participants will receive a weekly produce voucher redeemable at a local market vendor for fresh produce of the participant's choice. Participants will also receive a daily text message aimed to support a healthy diet and lifestyle. These texts will include information to build participants' knowledge and skills for healthy eating. The participants will also include weekly goals that focus on eating a healthy diet. Participants will receive automated, personalized feedback via text messages based on goal attainment and daily responses.
  Arms: Produce Voucher

SUMMARY:
The goal of this study is to understand the best practices for implementing produce prescriptions among adults with overweight or obesity experiencing nutrition insecurity. Enrolled participants will receive an 8-week intervention aimed at increasing nutrition knowledge, self-efficacy for healthy eating, and barriers to healthy food access. Participants will be randomly assigned to one of two produce prescription implementation strategies:

Program 1: Participants will receive weekly produce vouchers that are redeemable at a local vendor.

Program 2. Participants will receive fresh produce delivered directly to the participant's home. These boxes will be tailored based on household size, cooking and preparation preferences, and produce the participant prefers to receive.

Researchers will compare engagement in and adherence to the intervention and the patterns of difference in 8-week changes in fruit and vegetable consumption and weight.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 years of age or older
* Living with overweight or obesity, defined as a BMI ≥25
* Screens positive for nutrition insecurity
* Has a smartphone with a data plan
* Willing to receive daily text messages
* Has an address that can receive delivery
* Can read and write in English
* Is willing to pick up produce at the Northeast Market

Exclusion Criteria:

* Participating in another related research study
* Currently taking weight loss drugs
* Cardiovascular disease event in the last 6 months
* Active cancer
* Recent hospitalization due to psychiatric condition or event
* Pregnancy or planned during the study period
* Currently breastfeeding
* Documented dementia
* On kidney dialysis
* Planned or recent bariatric surgery
* Weight exceeding 440 lbs.
* Exclusion at principal investigators discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2025-01-08 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-06-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants Reached | 8 weeks
  The investigators will track the number of referrals, number of screening completions, number of eligible participants, and number of randomized participants, in addition to number of participants retained.

SECONDARY OUTCOMES:
Nutrition insecurity as assessed by the 4-item Nutrition Security Screening Questionnaire | Baseline, 4 weeks, 8 weeks
  Nutrition insecurity will be assessed using Center for Nutrition Health and Impact questionnaire with a 4-item scale that has a score range of 0-16. The higher the score, the greater the level of food security and control an individual has over their nutrition.
Change in Fruit and Vegetable Consumption as assessed by the 9-item Mini-Eating Assessment Tool (EAT) | Baseline, 4 weeks, and 8 weeks
  Consumption of food groups will be assessed using the 9-item Mini-Eating Assessment Tool (EAT) questionnaire. Each food group is assessed using a 9-point Likert scale ranging from I do not eat it at all to 6 or more servings per day. The survey is scored from 0-90 where a higher score indicates a healthier diet and a better outcome.
Weight (kg) | Baseline, 8 weeks
  Weight will be taken by study staff and measured to the nearest 0.1 kg.

CONTACTS AND LOCATIONS:
Overall Officials: Hailey Miller Assistant Professor, RN, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Northeast Market, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No